CLINICAL TRIAL: NCT05657678
Title: Efficacy Comparison of Two Doses of Vitamin D3 in Critically Ill Patients Undergoing Continuous Renal Replacement Therapy
Brief Title: Vitamin D3 Supplementation in Critically Ill Patients Undergoing CRRT
Acronym: NephroD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Tomasz Czarnik, MD PhD, Associate Professor, Uniwersytecki Szpital Kliniczny w Opolu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NephroD_2021
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Vitamin D3 Deficiency
Keywords: vitamin D; severe deficiency; continuous renal replacement therapy; intensive care; supplementation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Experimental): a single administration of 750,000 IU of vitamin D3 via the enteral route (through a gastric tube) in ICU patients with severe vitamin D3 deficiency (measured plasma 25(OH)D3 levels ≤12.5 ng/ml) undergoing continuous renal replacement therapy with CVVHDF or CVVHF
  Interventions: Drug: Vitamin D3 - 750 000 IU
- Control Arm (Active Comparator): a single administration of 500,000 IU of vitamin D3 via the enteral route (through a gastric tube) in ICU patients with severe vitamin D3 deficiency (measured plasma 25(OH)D3 levels ≤12.5 ng/ml) undergoing continuous renal replacement therapy with CVVHDF or CVVHF
  Interventions: Drug: Vitamin D3 - 500 000 IU

INTERVENTIONS:
Drug: Vitamin D3 - 750 000 IU — a single administration of 750,000 IU of vitamin D3
  Arms: Interventional Arm
Drug: Vitamin D3 - 500 000 IU — a single administration of 500,000 IU of vitamin D3
  Arms: Control Arm

SUMMARY:
Patients hospitalized in intensive care units (ICU) are particularly susceptible to vitamin D3 deficiencies. This can be due to the severity of their underlying disease, the type of treatment they are on, malnutrition before and inadequate nutrition during the hospitalisation preceding ICU admission, as well as advanced age. It has also been established that plasma levels of 25(OH)D3 tend to systematically decrease during ICU treatment. Therapeutic interventions administered in ICU settings such as fluid resuscitation or extracorporeal therapies can cause additional vitamin D3 deficiencies. The incidence of deficiency in critically ill patients can reach up to 90%, and even 30% of ICU patients can have undetectable plasma levels. It is impossible to replenish vitamin D3 levels in critically ill patients with traditional enteral and parenteral nutrition treatment regimens, because nutritional products contain too little of the vitamin. Vitamin D3 deficiency in critically ill patients has been associated with acute kidney injury, acute respiratory failure, sepsis, septic shock and increased all-cause ICU mortality. Despite that, assessment of plasma 25(OH)D3 levels is not a routine practice in ICUs. In view of the prevalence of vitamin D3 deficiencies in ICU patients, rapid replenishment of this deficiency with an increased supplementation dose should be considered as a potential means to improve prognosis in this patient population. The current standard therapy is the administration of 500,000 IU of vitamin D3 via the enteral route in ICU patients with severe deficiency (recommended by ESPEN). The NephroD study is meant to help answer the question whether increasing the standard ICU supplementation dose of vitamin D3 by 50% will ensure a more effective replenishment of this vitamin in critically ill patients undergoing CRRT.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of the following indications for initiation of CRRT with CVVHDF or CVVHF (acc. to KDIGO, Clinical Practice Guideline for Acute Kidney Injury):

   * replacement of kidney function in acute kidney injury
   * hyperkalaemia
   * metabolic acidosis
   * pulmonary oedema
   * uraemic complications (bleeding disorder, pericarditis)
   * hypervolaemia
   * support of renal function (volume control, regulation of acid-base and electrolyte status)
2. Sequential Organ Failure Assessment (SOFA) score of minimum 5 points at enrolment
3. Age of >18 years
4. Plasma 25(OH)D3 levels ≤12.5 ng/ml as measured by the local laboratory of a participating hospital
5. Properly managed enteral nutrition regardless of dosing

Exclusion Criteria:

1. Acute or advanced chronic liver failure (estimated on the basis of the clinical picture and biochemical markers: plasma bilirubin, plasma AST and ALT, high plasma AST/ALT ratio, glycaemia, INR)
2. Hypercalcaemia (total calcium concentration >11 mg/dl)
3. Any parathyroid disorder
4. End stage renal disease according to the KDIGO classification
5. Patients undergoing plasmapheresis, extracorporeal membrane oxygenation (ECMO), extracorporeal carbon dioxide removal (ECCO2R)
6. Patients who, in the opinion of the investigator, are not expected to survive 72 hours since enrolment
7. A history of nephrolithiasis or de novo nephrolithiasis
8. Patient qualified to a protocol for the avoidance of futile therapy
9. Pregnancy
10. Sarcoidosis
11. Risk of impaired intestinal absorption caused by the critical illness, associated with impaired peristalsis and delayed gastric emptying, constipation, diarrhoea, shock-induced intestinal hypoperfusion, hyperhydration with resulting intestinal oedema following fluid resuscitation, intestinal flora disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Supplementation | 7 days
  To evaluate and compare the effects of two different supplementation doses of vitamin D3 (25(OH)D3) - 500,000 IU or 750,000 IU administered as one enteral dose - on plasma levels of 25(OH)D3 in ICU patients undergoing continuous renal replacement therapy and diagnosed with severe vitamin D3 deficiency

SECONDARY OUTCOMES:
Mortality | 90 days
  To evaluate and compare the effects of two different supplementation doses of vitamin D3 on mortality in ICU patients undergoing continuous renal replacement therapy
ICU treatment duration | 90 days
  To evaluate and compare the effects of two different supplementation doses of vitamin D3 on ICU treatment duration in patients undergoing continuous renal replacement therapy
SOFA | 90 days
  To evaluate and compare the effects of two different supplementation doses of vitamin D3 on Sequential Organ Failure Assessment (SOFA) scores in ICU patients undergoing continuous renal replacement therapy
Catecholamines | 90 days
  To evaluate and compare the effects of two different supplementation doses of vitamin D3 on the duration of catecholamine administration in ICU patients undergoing continuous renal replacement therapy
CRRT | 7 days
  To evaluate the relationship between the length of CRRT use in hours from the time of study drug administration to the beginning of visit 4 and serum vitamin D3 levels in both study arms
GRV | 7 days
  To assess the relationship between total gastric residual volume (GRV) in millilitres from the time of study drug administration to the date of the beginning of visit 3 and serum vitamin D3 levels in both study arms

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Czarnik, MD, PhD, Principal Investigator — Uniwersytecki Szpital Kliniczny w Opolu
Locations (4):
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole, Opole Voivodeship
  - 5 Wojskowy Szpital Kliniczny z Poliklinika SP ZOZ, Krakow
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
  - Samodzielny Publiczny Szpital Kliniczny nr 1 Śląski Uniwersytet Medyczny w Katowicach, Zabrze

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Czarnik T, Bialka S, Borys M, Czuczwar M, Misiolek H, Piwowarczyk P, Szczeklik W, Wludarczyk A, Gawda R. Comparison of two doses of vitamin D3 in critically ill patients undergoing continuous renal replacement therapy (NephroD): study protocol for a single-blinded, multicenter, parallel group randomized controlled trial. Trials. 2024 Nov 24;25(1):791. doi: 10.1186/s13063-024-08598-5. PMID 39582029